CLINICAL TRIAL: NCT05177744
Title: An Innovative Analytical Platform to Investigate the Effect and Toxicity of Micro and Nano Plastics Combined With Environmental Contaminants on the Risk of Allergic Disease in Preclinical and Clinical Studies
Brief Title: Toxicity of Micro and Nano Plastics Combined With Environmental Contaminants on the Risk of Allergic Disease
Acronym: Imptox
Status: Completed | Type: Observational
Sponsor: Children's Hospital Srebrnjak (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Principal Investigator, Mirjana Turkalj, MD, Professor, MD, PhD, Children's Hospital Srebrnjak
Other Study IDs: SCH-EU965173
Record Dates: First submitted 2021-11-30; First posted 2022-01-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Food Hypersensitivity; Asthma in Children; Rhinitis, Allergic; Dermatitis, Atopic
MeSH Terms: conditions — Food Hypersensitivity; Rhinitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Whole blood and stool samples. Blood samples and stool samples will be collected twice (at baseline and after 6 months)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- allergic (Zagreb, urban): Participants will be selected based on proven sensitization to at least one food allergen (preferentially but not only to seafood) with a diagnosis of at least one allergic disease (i.e. allergic asthma, allergic rhinitis, atopic dermatitis and/or food allergy) for at least a year.
  Subjects will be recruited from continental region in Croatia - Zagreb (urban)
- healthy subjects (Zagreb, urban): Healthy subjects that will be recruited from continental region in Croatia - Zagreb (urban).
  Negative history of allergic diseases, as well as other severe chronic diseases, including malignant, autoimmune, or mental illnesses.
- allergic (Slavonia, urban and rural): Participants will be selected based on proven sensitization to at least one food allergen (preferentially but not only to seafood) with a diagnosis of at least one allergic disease (i.e. allergic asthma, allergic rhinitis, atopic dermatitis and/or food allergy) for at least a year.
  Subjects will be recruited from continental region in Croatia - Slavonia (urban and rural)
- healthy subjects (Slavonia, urban and rural): Healthy subjects that will be recruited from continental region in Croatia -(Slavonia, urban and rural).
  Negative history of allergic diseases, as well as other severe chronic diseases, including malignant, autoimmune, or mental illnesses.
- allergic Mediterranean region (urban and rural population): Participants will be selected based on proven sensitization to at least one food allergen (preferentially but not only to seafood) with a diagnosis of at least one allergic disease (i.e. allergic asthma, allergic rhinitis, atopic dermatitis and/or food allergy) for at least a year.
  Subjects will be recruited from mediterranean region in Croatia - urban and rural
- healthy subjects Mediterranean region (urban and rural population): Healthy subjects that will be recruited from mediterranean region in Croatia -urban and rural.
  Negative history of allergic diseases, as well as other severe chronic diseases, including malignant, autoimmune, or mental illnesses.

SUMMARY:
Single-center, cross-sectional, longitudinal, observational, population based cohort study with stratified sample (by age group, gender, and residential area).

DETAILED DESCRIPTION:
This study will involve schoolchildren (aged 6-18 years), population cohort based on differential exposure and susceptibility to allergy(paediatric population, allergic vs. healthy subjects). participants will be selected based on proven sensitization to at least one food allergen (preferentially but not only to seafood) with a diagnosis of at least one allergic disease (i.e. allergic asthma, allergic rhinitis (AR), atopic dermatitis (AD) and/or food allergy) for at least a year. Subjects will be recruited from three distinct and different geographical regions in Croatia: 2 continental regions (Zagreb, urban) and Slavonia (urban and rural) and 1 Mediterranean region (urban and rural population), differing in the levels of exposure (allergens, pollutants), consumption of water (main water source- bottled water, public water source, well water), food consumption (food packed in plastic material, use of fertilizers in agriculture), nutrition (food from marine environments, industrially processed food, homegrown food) as well as different environmental protection measures and human activities.In each region and subgroup, we will recruit 70 allergic children and 140 healthy (non-allergic) children in a cross-sectionalstudy protocol, summing up to al total of 630 participants.

The study will include visits:

1. Initial (screening) visit (V0 +3-6 months): written consent, assessment of inclusion and exclusion criteria, spirometry, Fractional exhaled nitric oxide (FeNO), questionnaires…
2. V2 (V0+6-9 months), questionnaires, environmental skin prick test (APT), sIgE (+ISAC), spirometry, FeNO, blood collection stool,
3. V2-V5 (V0+months 6-30 months)- regular visits (assessment) every 6 months, stool samples (second sampling)
4. Visit 4 (V0+18-24 months): environmental assessments, skin prick test (APT), sIgE (+ISAC), spirometry, FeNO, blood collection
5. V5 (last visit, V0+24-30 months)- final assessment of the study outcome measures, check and document consumption, adherence, preventive measures, level of control, therapy correction

Participants in the control group will be involved in collaboration with other outpatient clinics (eg. from surgical outpatient clinics who have had minor surgical procedures, from the Otorhinolaryngology- Ear, Nose, Throat (ENT) outpatient clinics at least 7 days after acute ear inflammation or laryngitis, from emergency ambulatory patients at least 7 days after acute respiratory illness, etc.). All participants who will be included in the control group should have a negative history of allergic diseases, as well as other severe chronic diseases, including malignant, autoimmune, or mental illnesses. They will need to fulfil the ISAAC questionnaire for children perform spirometry and prick test with a standard palette of inhalational and nutritional allergens to exclude allergic diseases.

No intervention tests or methods will be involved in this study. Patients who will be involved in the study will continue to take their regular therapy (according to guidelines) i.e. conduct treatment and all other non-therapeutic measures as if they were not involved in the study. Any deterioration or emergency intervention will be specifically evaluated and recorded as additional visits.

ELIGIBILITY:
Inclusion Criteria:

* Proven sensitization to at least one food allergen with a diagnosis of at least one allergic disease for at least one year
* Clinical diagnosis of allergic rhinitis (AR) for at least 1 year with symptoms of the nose, induced after exposure to allergens via IgE-mediated hypersensitivity reactions (symptoms of watery rhinorrhea, nasal obstruction, nasal itching and sneezing).
* Diagnosis of atopic dermatitis (AD) with AD symptoms lasting for more than 3 months, with or without food allergy

Additional inclusion criteria:

• Significant clinical allergy to indoor and outdoor allergens, an food allergens with positive skin prick test (SPT) and specific IgE levels (>0.35kUA/L)

Exclusion Criteria:

* Known inborn or perinatal pulmonary disease;
* Pulmonary malformation
* Oxygen therapy after birth with a duration of more than 24 h
* Ventilator support or mechanical ventilation after birth
* Diagnosis of cystic fibrosis
* Primary ciliary dyskinesia
* Heart failure diagnosed after birth affecting pulmonary circulation
* Major respiratory diseases such as e.g. interstitial lung disease and other congenital and serious chronic disease
* Fever of at least 38.5 °C during the last two weeks prior to the planned visit

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants in the control group will be involved in collaboration with other outpatient clinics (eg. from surgical outpatient clinics who have had minor surgical procedures, from the ENT outpatient clinics at least 7 days after acute ear inflammation or laryngitis, from emergency ambulatory patients at least 7 days after acute respiratory illness, etc.). All participants who will be included in the control group should have a negative history of allergic diseases, as well as other severe chronic diseases, including malignant, autoimmune, or mental illnesses.
Sampling Method: Probability Sample
Enrollment: 1156 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Lung function tests | 6 months, Asthmatic patients will be regularly controlled even more often in case of exacerbations.
  Forced expiratory volume in one second (FEV1), Forced vital capacity (FVC) and the ratio of the two volumes (FEV1/FVC) will be recorded for each patient at each visit.
  FEV1 is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration. It's measured in % of predicted values which are the average readings that would be expected in a healthy person of similar age, gender, body size, and ethnicity.
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, measured in liters.

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide (FeNO) | 6 months, Asthmatic patients will be regularly controlled even more often in case of exacerbations
  FeNO test measures the level of nitric oxide gas in an exhaled sample of breath. It is measured in "parts per billion" (ppb).
Childhood Asthma Control Test (C-ACT) | 6 months, Asthmatic patients will be regularly controlled even more often in case of exacerbations
  C-ACT questionnaire will be used to tell us if the asthma treatment plan is optimal and if asthma is being properly controlled. For children 4 to 11 years maximal score is 27, and for those older then 12 years maximal score is 25. Higher scores reflect greater asthma control, and if the score is 19 or less may be a sign that asthma is not controlled as well as it could be.
Daily burden of disease (Global evaluation) | 6 months, Asthmatic patients will be regularly controlled even more often in case of exacerbations
  Participants' daily burden of disease will be evaluated by visual analogue scale (VAS) Visual analogue scale levels <20/100 were categorized as "Low" burden and VAS levels ≥50/100 as "High" burden.
Daily burden of disease (affecting Nose) | 6 months
  Participants with AR will be evaluated by visual analogue scale (VAS).Visual analogue scale levels <20/100 were categorized as "Low" burden and VAS levels ≥50/100 as "High" burden.
Daily burden of disease (affecting Eyes) | 6 months
  Participants' daily burden of the disease affecting eyes will be evaluated by visual analogue scale (VAS).Visual analogue scale levels <20/100 were categorized as "Low" burden and VAS levels ≥50/100 as "High" burden.
Daily burden of disease (Asthma) | 6 months, Asthmatic patients will be regularly controlled even more often in case of exacerbations
  Participants' daily burden of asthma will be evaluated by visual analogue scale (VAS).Visual analogue scale levels <20/100 were categorized as "Low" burden and VAS levels ≥50/100 as "High" burden.
SCORing Atopic Dermatitis (SCORAD) | 6 months for patients with AD
  SCORAD as a clinical tool will be used to assess the extent and severity of eczema. The SCORAD Index formula is: A/5 + 7B/2 + C. In this formula A is defined as the extent (0- 100), B is defined as the intensity (0- 18) and C is defined as the subjective symptoms (0- 20). The maximal score of the SCORAD Index is 103.

OTHER OUTCOMES:
ISAC platform | Blood samples will be collected twice (at baseline and after 6 months)
  Detailed assessment of allergic sensitization will be performed using ISAC platform with the analysis of >100 allergic components of food and/or inhalatory allergens. Serum concentrations of the specific IgEs reacting to 103 allergen components from 43 allergen sources will be measured using the Multiplex Component Diagnosis (ISAC) platform. ISAC is a semi-quantitative test and results are reported in ISAC standard units (ISU) indicating specific IgE-antibody levels; the operating range is 0.3-100 ISU-E. This range is about the same as a concentration range of 0.3-100 kilo international units of allergen-specific antibody per unit volume of sample (kUA/litre) of IgE (1 kUA/litre is equal to 2.4 nanograms/ml).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, City of Zagreb, Croatia